CLINICAL TRIAL: NCT02521974
Title: A Phase 4 Study to Evaluate the Safety and Immunogenicity of Monovalent Oral Polio Vaccine Type 2 in Healthy Children Aged 1 to 5 Years and in bOPV-IPV Vaccinated Healthy Infants
Brief Title: A Study to Evaluate the Safety and Immunogenicity of Oral Polio Vaccine Type 2 in Infants and Children
Acronym: M2-ABMG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fidec Corporation (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: M2-ABMG
Record Dates: First submitted 2015-07-31; First posted 2015-08-13 (Estimated); Results first posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2017-07

CONDITIONS: Adverse Event Following Immunisation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SABIN monovalent OPV2 vaccine (Experimental): SABIN monovalent OPV2 is a licensed, monovalent, live attenuated poliomyelitis virus vaccine of the Sabin strain Type 2 (P 712, Ch, 2ab), propagated in MRC5 human diploid
  Interventions: Biological: SABIN monovalent OPV2

INTERVENTIONS:
Biological: SABIN monovalent OPV2 — SABIN monovalent OPV2 is a licensed, monovalent, live attenuated poliomyelitis virus vaccine of the Sabin strain Type 2 (P 712, Ch, 2ab), propagated in MRC5 human diploid cells. Each two-drop dose (0.1 mL) contains not less than 105.0 CCID50 of Type 2
  Other Names: Polio Sabin™ Mono Two (oral)

SUMMARY:
Sabin 2 will be withdrawn from routine use globally from April 2016 as per the SAGE recommendations at the time of writing this protocol. After this cessation of OPV2, stockpiles of mOPV2 will be maintained for potential use if necessary in response to a future outbreak. However, there will be a risk of cVDPV2 from Sabin 2 in settings of low population immunity. Research is ongoing to develop vaccines that are genetically more stable than the currently available Sabin 2-containing OPVs. To generate data on immunogenicity, safety, and genetic stability on the Sabin 2 vaccine (mOPV2) and as a future comparator for new polio vaccine research after the global switch from tOPV to bOPV, this study with mOPV2 is performed to evaluate safety, immunogenicity (humoral and intestinal) and genetic stability endpoints of mOPV2 in children aged 1 to 5 years and in infants approximately 18 weeks of aged vaccinated with bOPV-/IPV for better understanding of the stockpile use of this vaccine, and for comparison with any potential new polio vaccine with a type 2 component in the future.

DETAILED DESCRIPTION:
1. PRIMARY OBJECTIVE The primary objectives of the study are to assess the safety (serious adverse events [SAEs] and severe adverse events [AEs] grade 3 according to CTCAE 4.03 and immunogenicity (seroprotection rate) of a single dose of SABIN mOPV2 in healthy children aged 1 to 5 years old, and in infants at approximately 18 weeks of age after having been vaccinated with 3 doses of bOPV and 1 dose of IPV .
2. SECONDARY OBJECTIVES

   Secondary objectives are to assess:
   * The safety (mild and moderate solicited and unsolicited AEs, Important Medical Events [IMEs], and laboratory deviation assessments) of one or two doses of SABIN mOPV2 in healthy children aged 1 to 5 years, and of 2 doses of SABIN mOPV2 in infants at approximately 18 and 22 weeks of age after having been vaccinated with 3 doses of bOPV and 1 dose of IPV.
   * The immunogenicity (seroconversion rate, median and geometric mean antibody titers) of one or two doses of SABIN mOPV2 in healthy children aged 1 to 5 years old, and of two doses of SABIN mOPV2 in infants at approximately 18 22 weeks of age after having been vaccinated with 3 doses of bOPV and 1 dose of IPV.
3. EXPLORATORY OBJECTIVES

Exploratory objectives are:

* To investigate viral shedding following the SABIN mOPV2 administration.
* Exploratory objectives may also include assessment of the genetic sequence heterogeneity and potential for neurovirulence (as measured in animal model(s)) of shed virus.
* To investigate viral shedding and neurovirulence of shed virus;
* To evaluate genetic reversion at position nt481 (primarily) and other secondary sites (e.g., nt2908).
* To investigate the priming responses of bOPV for mOPV2. (group 2 only) and the duration of induction of anti-polio type 2 neutralizing antibodies .

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 1 to 5 years previously vaccinated with three or four doses of IPV (Group 1) or unvaccinated infants aged 6 weeks (-7 to +14 days) (Groups 2 and 3).
2. For Groups 2 and 3 (enrolled at 6 weeks of age) infants must have been vaccinated with 3 doses of bOPV and one dose of IPV prior to administration of the study vaccine, and the last Polio vaccine must have been administered at least 4 weeks prior to the study vaccine.
3. Healthy without obvious medical conditions that preclude the subject to be in the study as established by the medical history and physical examination.
4. Written informed consent obtained from 1 or 2 parent(s) or legal guardian(s) as per country regulations.

Exclusion Criteria:

1. For Group 1: polio vaccines within the 3 months prior to the administration of the study vaccine (number of previous polio vaccine doses to be documented). For Groups 2 and 3: polio vaccines prior to administration of the study vaccine other than 3 doses of bOPV and 1 dose of IPV .
2. Any confirmed or suspected immunosuppressive or known immunodeficient condition including human immunodeficiency virus (HIV) infection.
3. Family history of congenital or hereditary immunodeficiency.
4. Major congenital defects or serious uncontrolled chronic illness (neurologic, pulmonary, gastrointestinal, hepatic, renal, or endocrine).
5. Known allergy to any component of the study vaccines or to any antibiotics.
6. Uncontrolled coagulopathy or blood disorder contraindicating intramuscular injections (of IPV).
7. Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
8. Acute severe febrile illness at day of vaccination deemed by the Investigator to be a contraindication for vaccination (the child can be included at a later time if within age window and all in/exclusion criteria are met.).
9. Member of the subject's household (living in the same house or apartment unit) has received OPV in the last 3 months.
10. Subject who, in the opinion of the Investigator, is unlikely to comply with the protocol or is inappropriate to be included in the study for the safety or the benefit-risk ratio of the subject.

Ages: 6 Weeks to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 164 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier M Saez-Llorens, MD, Principal Investigator — Hospital del Niño de Panama

REFERENCES:
- [Derived] Wahid R, Mercer LD, De Leon T, DeAntonio R, Saez-Llorens X, Macadam A, Chumakov K, Strating J, Koel B, Konopka-Anstadt JL, Oberste MS, Burns CC, Andino R, Tritama E, Bandyopadhyay AS, Aguirre G, Ruttimann R, Gast C, Konz JO. Genetic and phenotypic stability of poliovirus shed from infants who received novel type 2 or Sabin type 2 oral poliovirus vaccines in Panama: an analysis of two clinical trials. Lancet Microbe. 2022 Dec;3(12):e912-e921. doi: 10.1016/S2666-5247(22)00254-3. Epub 2022 Nov 1. PMID 36332645
- [Derived] Saez-Llorens X, Bandyopadhyay AS, Gast C, Leon T, DeAntonio R, Jimeno J, Caballero MI, Aguirre G, Oberste MS, Weldon WC, Konopka-Anstadt JL, Modlin J, Bachtiar NS, Fix A, Konz J, Clemens R, Costa Clemens SA, Ruttimann R. Safety and immunogenicity of two novel type 2 oral poliovirus vaccine candidates compared with a monovalent type 2 oral poliovirus vaccine in children and infants: two clinical trials. Lancet. 2021 Jan 2;397(10268):27-38. doi: 10.1016/S0140-6736(20)32540-X. Epub 2020 Dec 9. PMID 33308427

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: 1-5 years old children who had previously been fully vaccinated with OPV and/or IPV and who will received 2 doses of the investigational vaccine.
- Group 2+3: 18 - 22 weeks old infants who will first receive bOPV/IPV coverage and one / two dose / s of the investigational vaccine.
Period: Overall Study
Arm/Group | Group 1 | Group 2+3
Started | 50 | 114
Completed | 47 | 110
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Population: 4 early terminated subjects during the pre-vaccination phase, before receiving the investigational vaccine.
Groups:
- Group 2+3: 18 - 22 weeks old infants who will first receive bOPV/IPV coverage and one / two dose/s of the investigational vaccine.
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2+3 | Total
Number analyzed (Participants) | 50 | 110 | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 50 | 110 | 160
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 49 | 78
  Male | 21 | 61 | 82
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 50 | 110 | 160
Region of Enrollment [Count of Participants; unit: Participants]
  Panama | 50 | 110 | 160

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Experiencing SAEs, Severe AEs (Grade 3), and/or IMEs
Description: Number of subjects experiencing SAEs, severe AEs (grade 3), and IMEs considered consistent with a causal association to study vaccine throughout the study period in all groups.
Time Frame: 6 months
Population: 50 (100%) children in Group 1 received the first dose of study vaccine and 47 (94%) children received the second dose. All 110 (100%) infants in combined Groups 2+3 received the first dose of study vaccine and 49 (98.0%) of the 50 infants in Group 3 received 2 doses of vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2+3
Number analyzed (Participants) | 50 | 110
Participants | 0 | 1

2. Primary Outcome: Seroprotection Rate of Type 2 Polio Neutralizing Antibodies.
Description: Measured at Day 28 following a single dose of Sabin mOPV2 in both infant groups (Groups 2+3).
  Seroprotection is defined as type 2-specific antibody titers ≥1:8 and seroprotection rate as the percentage of seroprotected subjects per group.
Time Frame: 28 days
Population: TVP is 110 while PP is 97 - per protocol the PP population will be used for immunogenicity analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2+3
Number analyzed (Participants) | 97
Participants | 91

ADVERSE EVENTS:
Arm/Group | Group 1 | Group 2+3
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/114
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/114
Other Adverse Events (participants affected / at risk) | 1/50 | 1/114
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=50) | Group 2+3 (N=114)
Abnormal crying (General disorders) | 0 | 1
Irritability (General disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No